CLINICAL TRIAL: NCT00726544
Title: A Randomized, Double-blind, Placebo Controlled, Clinical Outcome Study of ARC1779 Injection in Patients With Thrombotic Microangiopathy
Brief Title: Clinical Outcome Study of ARC1779 Injection in Patients With Thrombotic Microangiopathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment into study was slower than expected.
Sponsor: Archemix Corp. (Industry)
Responsible Party: Dr, James Gilbert, Archemix
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARC1779-006
Record Dates: First submitted 2008-07-30; First posted 2008-08-01 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2009-11

CONDITIONS: Thrombotic Microangiopathy; Thrombotic Thrombocytopenic Purpura
Keywords: thrombocytopenia; microangiopathic hemolytic anemia; von Willebrand Factor; ADAMTS13
MeSH Terms: conditions — Thrombotic Microangiopathies; Purpura, Thrombotic Thrombocytopenic; Thrombocytopenia; Anemia, Hemolytic | interventions — ARC 1779

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: ARC 1779 Placebo
- Low Dose (Active Comparator)
  Interventions: Drug: ARC1779 Injection
- Medium Dose (Active Comparator)
  Interventions: Drug: ARC1779 Injection
- High Dose (Active Comparator)
  Interventions: Drug: ARC1779 Injection

INTERVENTIONS:
Drug: ARC 1779 Placebo — ARC1779 Injection or placebo is administered intravenously to patients as an initial loading dose followed by continuous infusion of up to 14 days plus 2 day taper.
  Arms: Placebo
Drug: ARC1779 Injection — ARC1779 Injection or placebo is administered intravenously to patients as an initial loading dose followed by continuous infusion of up to 14 days plus 2 day taper. Treatment with ARC1779 Injection is to be given at low dosage that is intended to produce target steady-state ARC1779 plasma concentrations during infusion of 3μg/mL.
  Arms: Low Dose
Drug: ARC1779 Injection — ARC1779 Injection or placebo is administered intravenously to patients as an initial loading dose followed by continuous infusion of up to 14 days plus 2 day taper. Treatment with ARC1779 Injection is to be given at low dosage that is intended to produce target steady-state ARC1779 plasma concentrations during infusion of 6μg/mL.
  Arms: Medium Dose
Drug: ARC1779 Injection — ARC1779 Injection or placebo is administered intravenously to patients as an initial loading dose followed by continuous infusion of up to 14 days plus 2 day taper. Treatment with ARC1779 Injection is to be given at low dosage that is intended to produce target steady-state ARC1779 plasma concentrations during infusion of 12μg/mL.
  Arms: High Dose

SUMMARY:
The purpose of this ascending-dose research study is to determine whether the administration of ARC1779 Injection improves subject's health profile by protecting the brain, heart, and kidney from damage due to formation of small blood clots in blood vessels. It will also determine the safety of ARC1779 Injection, how ARC1779 Injection enters and leaves the blood and tissue over time, and its effect on laboratory tests related to blood clotting, heart and brain function, and other body systems.

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* ≥18 to ≤75 years of age;
* Diagnosis of TMA based on presence of:
* Thrombocytopenia, defined as a platelet count <100 x 109 per liter;
* Microangiopathic hemolytic anemia, defined by negative findings on direct antiglobulin test, and evidence of accelerated red blood cell (RBC) production and destruction); AND
* Absence of a clinically apparent alternative explanation for thrombocytopenia and anemia, e.g., disseminated intravascular coagulation (DIC), eclampsia, HELLP syndrome, Evans syndrome;
* Females: non-pregnant and commit to use of effective, redundant methods of contraception (i.e., for both self and male partner) throughout the study and for at least 30 days after discontinuation of study drug treatment;
* Males: commit to use of a medically acceptable contraceptive (abstinence or use of a condom with spermicide) throughout the study and for at least 30 days after discontinuation of study drug treatment;
* Not received an unlicensed investigational agent (drug, device, or blood-derived product) within 30 days prior to randomization, and may not receive such an investigational agent in the 30 days post-randomization (note: investigational use for treatment of TMA of a licensed immunomodulator, e.g., rituximab, is permitted at any time relative to randomization);
* Capable of understanding and complying with the protocol, and he/she (or a legal representative) must have signed the informed consent document prior to performance of any study-related procedures.

Patients who have again become acutely ill following recent treatment and achievement of a brief remission of acute TMA may be enrolled in the study if ALL of the following conditions are met:

* Disease activity in the patient in unabated (e.g. persistent thrombocytopenia and microangiopathic hemolytic anemia with ongoing neurological symptoms and/or troponin elevation);
* The last plasma exchange of the patient's preceding course of treatment occurred at least 7 days prior;
* The patient did not undergo splenectomy during the preceding course of treatment;
* The new course of plasma exchange has not been ongoing for more than 3 days.

Exclusion Criteria:

* Females: pregnant or <24 hours post-partum, or breastfeeding;
* History of bleeding diathesis or evidence of active abnormal bleeding within the previous 30 days;
* Disseminated malignancy or other co-morbid illness limiting life expectancy to ≤3 months independent of the TMA disorder.
* Diagnosis other than TMA which can account for the findings of thrombocytopenia and hemolytic anemia (e.g., DIC, HELLP syndrome, Evans syndrome);
* Diagnosis of DIC verified by laboratory values for D-dimer, fibrinogen, prothrombin time (PT), and activated partial thromboplastin time (aPTT).

Patients who have again become acutely ill following recent treatment and achievement of a brief remission of acute TMA may not be enrolled in the study if ANY of the following conditions are met:

* The last plasma exchange of the patient's preceding course of treatment occurred less than 7 days prior;
* The patient underwent splenectomy during the preceding course of treatment;
* The new course of plasma exchange has been ongoing for more than 3 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-12; Primary Completion 2010-12 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
The incidence of the clinical composite of death (all-cause mortality), stroke, coma, seizures, renal failure, or acute myocardial infarction (AMI) | 6 weeks post randomization

SECONDARY OUTCOMES:
Neurocognitive function is to be assessed with the CogState® test system. | Once during the hospitalization period and again at the 6 week clinic visit.
The incidence of death, stroke, or acute renal failure/injury requiring dialysis is to be assessed. | During the extended clinical follow-up for each patient from the time of the 6 week clinic visit until the study is closed.
Safety- and efficacy-related clinical laboratory parameters and biomarkers will be analyzed in relation to ARC1779 exposure in terms of the dose administered and the observed plasma concentration. | During initial hospitalization and at 6 week clinic visit.
The incidence of the composite of complications associated with plasma exchange therapy (i.e., catheter-related infection, thrombosis, internal hemorrhage, or pneumothorax) is to be assessed. | During initial hospitalization and at the 6 week clinic visit.

CONTACTS AND LOCATIONS:
Locations (17):
- United States (7):
  - Northwestern University, Chicago, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Washington University, St Louis, Missouri
  - New York Medical College, Valhalla, New York
  - The Ohio State University Research Foundation, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - The Methodist Hospital, Houston, Texas
- University of Vienna, Vienna, Austria
- Canada (3):
  - QEII CDHA Centre, Halifax, Nova Scotia
  - CICM/Hospital Charles LeMoyne, Greenfield Park, Quebec
  - CHA-Hospital de L'Enfant-Jesus, Québec, Quebec
- Italy (5):
  - Ospedale Ferrarotto, Catania
  - Policlinico Mangiagalli Regina Elena-Fondazione L.Villa, Milan
  - Fondazione Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera S.Maria Nuova, Reggio Emilia
  - Università Cattolica del Sacro Cuore, Rome
- University College London Hospital, London, United Kingdom